CLINICAL TRIAL: NCT06317883
Title: Longitudinal Study To Determine The Risk Factors Associated With Childhood Obesity
Brief Title: Childhood Obesity Risk Assessment Longitudinal Study
Acronym: CORALS
Status: Active, not recruiting | Type: Observational
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government); Maimónides Biomedical Research Institute of Córdoba (Other); Universidad de Córdoba (Other); Institut Investigacio Sanitaria Pere Virgili (Other); University Rovira i Virgili (Other); Centro de Investigación Biomédica en Red de Fisiopatología de la Obesidad y Nutrición (CIBEROBN) (Unknown); Universidad de Zaragoza (Other); University of Valencia (Other); University of Navarra (Other); Hospital Clinico Universitario de Santiago (Other); University of Santiago de Compostela (Other); Health Research Institute of Santiago (Other); Hospital del Mar Research Institute (IMIM) (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Universidad de Granada (Other); Biosanitary Research Institute of Granada (Unknown)
Responsible Party: Sponsor
Other Study IDs: CORALS
Record Dates: First submitted 2024-02-07; First posted 2024-03-19 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Child Obesity
Keywords: Childhood obesity; Dietary pattern; Sedentary behaviors; Physical activity; Cardiometabolic risk factors
MeSH Terms: conditions — Pediatric Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood and stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CORALS: Children aged 3-6 years

SUMMARY:
Childhood obesity is a major public health problem worldwide. Europe has a high prevalence of obesity, which is accentuated in Mediterranean countries. Spain has a high prevalence of both overweight (percentage: 21.5 in boys and 22.2 in girls) and obesity (percentage: 10.6 in boys and 11.8 in girls) in children aged 6-9 years.

From childhood, obesity is associated with an increased risk of diseases such as insulin resistance, type 2 diabetes, hypertension, metabolic syndrome, musculoskeletal problems, sleep disorders and mental health problems. Obesity is a complex, multi-causal problem involving individual risk factors such as behavior and genetics. Behavioral factors include diet, physical activity, sedentary lifestyle, sleep, and others. It is therefore important to study each of the individual risk factors for obesity. There are few large sample studies in European/Spanish children and no longitudinal studies estimating the incidence of obesity in preschool children based on exposure to different risk factors, considering not only the effect of food consumption but also dietary habits and patterns.

The aim of the present study is to identify risk factors for childhood obesity through long-term longitudinal follow-up.

DETAILED DESCRIPTION:
This is a longitudinal, multi-centre prospective cohort study of children aged 3-6 years with annual data collection for an average follow-up of 10 years.

The main objective of the present study is to identify risk factors for childhood obesity through long-term longitudinal follow-up. At least 2,214 participants are required.

The specific objectives are as follows:

1. Assess the associations between perinatal risk factors, socioeconomic, cultural and environmental factors and the risk of developing obesity and its comorbidities.
2. Assess the associations between lifestyles (diet, beverage consumption, physical activity, sedentary lifestyle, sleep) and the risk of developing obesity and its comorbidities.
3. Evaluate the association between genetic polymorphisms, metabolomic and metagenomic profiles (determined by omics techniques) and the development of obesity and its comorbidities.

Study design

The selection visit includes:

A) The administration of a face-to-face questionnaire to check eligibility criteria. Only if the participant is eligible the screening visit will proceed to b).

B) Explanation and clarification of any doubts about the study, delivery of the study information sheet to the participant and completion of the informed consent form signed by both parents (essential for inclusion in the study).

C) The family will be provided with a 3-day prospective food record (2 working days and 1 weekend day), the general data collection booklet and the following questionnaires: adherence of the primary tutor to the Mediterranean diet, dietary behavior, psychosocial, active lifestyle, sedentary behavior and sleep patterns. These questionnaires are to be returned at the next visit.

D) Instructions and bottles for collecting biological samples are given.

Inclusion visit includes:

1. Review of the 3-day food record and all questionnaires from the selection visit.
2. Once the inclusion and exclusion criteria have been evaluated, the participant will be included in the study if all the requirements are met. Then, the next step will be taken.
3. Completion of the 14-point Mediterranean diet adherence questionnaire (to be completed by the primary tutor), baseline questionnaire (height, weight, waist, bioimpedance, blood pressure, child's active lifestyle and Mediterranean diet adherence) and the food and drink frequency questionnaire.
4. Performing a speech fluency test and a fitness assessment examination.
5. Collection of blood, urine, and stools samples.
6. If the participant has an odd-numbered ID, an accelerometer is provided to be used for 7 consecutive days. Collected data must be recorded in a diary.

After the inclusion visit, the participant will undergo two types of follow-up visits in which the following evaluations will be made:

Follow-up visits - Years 01, 02, 04, 06, 07, 08 and 09

1. Baseline questionnaire without collecting biological samples
2. Food frequency questionnaire
3. 14-point Mediterranean diet adherence questionnaire

Follow-up visits - Years 03, 05 and 10 Completion of all questionnaires and determinations corresponding to the inclusion visit.

A window of ±3 months of the corresponding follow-up year since the inclusion visit is allowed.

Justification: The results of this study could help to understand and act on the key determinant factors of the epidemic of overweight and obesity in children.

Long-term follow-up of a large cohort is necessary to develop strategies to combat the serious consequences that overweight and obesity cause on the spanish public health system. This is an important objective and a clear public health priority, since it addresses both the main epidemic of our time (childhood overweight/obesity) as the main cause of healthcare expenditure at increasingly younger ages that makes the current healthcare system unviable (chronic diseases).

The project involves a large number of children from early childhood and follows them over time, covering the key ages for the establishment of dietary habits, lifestyles and adipose rebound. The study can allow the transfer and translation to the general population and the integration of epidemiological, clinical and basic aspects in the proposed research.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 6 years.
* Compliance with the 3-day food consumption record, the free time physical activity questionnaire and attendance at the scheduled inclusion visit together with the delivery of the signed informed consent.

Exclusion Criteria:

* Children from families with difficulties in participating or complying with the study protocol, as well as difficulties with comprehension, language, or unstable domicile.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3-6 years.
Sampling Method: Probability Sample
Enrollment: 1508 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2032-07-14 (Estimated); Study Completion 2032-07-14 (Estimated)

PRIMARY OUTCOMES:
Assessment of dietary intake and habits | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  The habitual intake of the child is assessed by using the food and drink frequency questionnaire and the 14-point Mediterranean diet adherence questionnaire. In addition, a food behaviour questionnaire is administered to the child's parents or primary caregiver.
Assessment of physical activity, sedentary behavior and sleep pattern | 0, 3, 5 and 10 years since the selection visit.
  Sedentary activities are assessed by means of an ad hoc questionnaire on the time children spend watching television, using computers, cell phones, video games and consoles, as well as their sleep patterns. Likewise, physical activity is assessed by (1) an ad hoc questionnaire to determine the active lifestyle of the children and (2) an accelerometries (half of the participants).
Early risk factors | 0, 3, 5 and 10 years since the selection visit.
  The parents of the children are asked to fill out a general questionnaire that request information regarding: personal and family history related to pregnancy, diseases, lifestyle, toxic habits, weight gain, lifestyle, toxic habits, and others.
Body composition: Height | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Height in centimeters is measured with the SECA 213 precision measuring instrument on an annual basis.
Body composition: Weight | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Weight in grams is measured by the precision weighing scale model Tanita 780PMA on an annual basis.
Body composition: Body mass index | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Body mass index in kilograms per square meter is calculated on an annual basis.
Body composition: Waist circumference | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Waist circumference in centimeters is measured with a SECA 201 precision measuring tape on an annual basis.
Psychosocial and neuropsychological behavioral assessment | 0, 3, 5 and 10 years since the selection visit.
  Strengths and Difficulties Questionnaire (SDQ), an internationally recognized and validated questionnaire is used to assess the general behavior. The questionnaire is to be answered by the parents/tutor on an individual basis, focusing on the behavior of his/her son/daughter during the last 6 months. This questionnaire covers emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior.
  The SDQ contains 5 subscales (4 dysadaptive and 1 adaptive [prosocial scale]). Each has a range of 0 to 10 points. The SDQ score range is 0-40 points (excluding the prosocial scale), with 0 being considered normality.
Verbal fluency | 0, 3, 5 and 10 years since the selection visit.
  Normative data from phonological and semantic verbal fluency tests (VFT) in Spanish-speaking pediatric populations is followed to assess verbal fluency, one of the most sensitive indicators of cognitive development, especially executive function.
Muscular strength | 0, 3, 5 and 10 years since the selection visit.
  Muscle strength is assessed by measuring both hand grip strength in kilograms and lower body explosive strength - a long jump with the feet together- in centimeters.
Cardiorespiratory endurance | 0, 3, 5 and 10 years since the selection visit.
  Cardiorespiratory endurance is assessed in minutes by using the Course Navette test. The number of completed series is recorded.

SECONDARY OUTCOMES:
Association between genetic polymorphisms, metabolomic and metagenomic profiles with the development of obesity. | 0, 3, 5 and 10 years since the selection visit.
  Aliquots of plasma, serum, and leukocyte layer are to be stored for DNA isolation for genetic/epigenetic analysis to investigate genetic, metabolomic, and epigenetic associations with the development of obesity.
Body composition: Waist height | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Waist height in centimeters is measured on an annual basis.
Body composition: Fat mass | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Fat mass both in kilograms and in percentage is measured on an annual basis.
Body composition: Fat mass index | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Fat mass index in kilograms per square meter is calculated on an annual basis.
Body composition: Fat-free mass | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Fat-free mass in kilograms is measured on an annual basis.
Body composition: Total body water | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  Total body water both in kilograms and in percentage is measured on an annual basis.
Systolic blood pressure measurement | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  On an annual basis, the systolic blood pressure is measured in mmHg in triplicate in order to obtain an average value.
Diastolic blood pressure measurement | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  On an annual basis, the diastolic blood pressure is measured in mmHg in triplicate in order to obtain an average value.
Heart rate measurement | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 years since the selection visit.
  On an annual basis, the heart rate is measured in beats per minute in triplicate in order to obtain an average value.
Hematological analysis: Hemoglobine | 0, 3, 5 and 10 years since the selection visit.
  Hemoglobin levels are determined in grams per deciliter on an individual basis.
Hematological analysis: Hematocrite | 0, 3, 5 and 10 years since the selection visit.
  Hematocrite levels are determined in percentage on an individual basis.
Hematological analysis: Erythrocytes | 0, 3, 5 and 10 years since the selection visit.
  Erythrocytes count is measured in 10e06 units per microliter on an individual basis.
Hematological analysis: Mean corpuscular volume | 0, 3, 5 and 10 years since the selection visit.
  Mean corpuscular volume is measured in femtoliters on an individual basis.
Hematological analysis: Mean corpuscular hemoglobin | 0, 3, 5 and 10 years since the selection visit.
  Mean corpuscular hemoglobine is measured in picograms on an individual basis.
Hematological analysis: Mean corpuscular hemoglobin concentration | 0, 3, 5 and 10 years since the selection visit.
  Mean corpuscular hemoglobine concentration is measured in grams per deciliter on an individual basis.
Hematological analysis: Red cell blood distribution width | 0, 3, 5 and 10 years since the selection visit.
  Red cell blood distribution width is determined in percentage on an individual basis.
Hematological analysis: White blood cells | 0, 3, 5 and 10 years since the selection visit.
  White blood cells count is measured in 10e03 units per microliter on an individual basis.
Hematological analysis: Neutrophils | 0, 3, 5 and 10 years since the selection visit.
  Neutrophils count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Lymphocytes | 0, 3, 5 and 10 years since the selection visit.
  Lymphocytes count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Monocytes | 0, 3, 5 and 10 years since the selection visit.
  Monocytes count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Eosinophils | 0, 3, 5 and 10 years since the selection visit.
  Eosinophils count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Basophiles | 0, 3, 5 and 10 years since the selection visit.
  Basophiles count is measured both in 10e03 units per microliter and in percentage on an individual basis.
Hematological analysis: Platelets | 0, 3, 5 and 10 years since the selection visit.
  Platelets count is measured in 10e03 units per microliter on an individual basis.
Hematological analysis: Mean platelet volume | 0, 3, 5 and 10 years since the selection visit.
  Mean platelet volume is measured in femtoliters on an individual basis.
Biochemical analysis: Glucose | 0, 3, 5 and 10 years since the selection visit.
  Glucose is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Bilirubin | 0, 3, 5 and 10 years since the selection visit.
  Total bilirubin is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Creatinine | 0, 3, 5 and 10 years since the selection visit.
  Creatinine is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Urate | 0, 3, 5 and 10 years since the selection visit.
  Urate is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Urea | 0, 3, 5 and 10 years since the selection visit.
  Urea is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total protein | 0, 3, 5 and 10 years since the selection visit.
  Total protein is measured both in grams per deciliter and in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Aspartate aminotransferase | 0, 3, 5 and 10 years since the selection visit.
  Aspartate aminotransferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Alanine aminotransferase | 0, 3, 5 and 10 years since the selection visit.
  Alanine aminotransferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Gamma-glutamyl transferase | 0, 3, 5 and 10 years since the selection visit.
  Gamma-glutamyl transferase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Alkaline phosphatase | 0, 3, 5 and 10 years since the selection visit.
  Alkaline phosphatase is measured in international units per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total cholesterol | 0, 3, 5 and 10 years since the selection visit.
  Total cholesterol is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: High density lipoproteins | 0, 3, 5 and 10 years since the selection visit.
  High density lipoproteins (HDL) are measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Non-HDL cholesterol | 0, 3, 5 and 10 years since the selection visit.
  Non-HDL cholesterol levels are calculated in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Low density lipoproteins | 0, 3, 5 and 10 years since the selection visit.
  Low density lipoproteins (LDL) are measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Apolipoprotein A1 | 0, 3, 5 and 10 years since the selection visit.
  Apolipoprotein A1 is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Apolipoprotein B | 0, 3, 5 and 10 years since the selection visit.
  Apolipoprotein B is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Calcium | 0, 3, 5 and 10 years since the selection visit.
  Calcium is measured both in milligrams per deciliter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Potassium | 0, 3, 5 and 10 years since the selection visit.
  Potassium is measured both in millimoles per liter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Sodium | 0, 3, 5 and 10 years since the selection visit.
  Sodium is measured in millimoles per liter, in milliequivalents per liter and in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Phosphorus | 0, 3, 5 and 10 years since the selection visit.
  Phosphorus is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Iron | 0, 3, 5 and 10 years since the selection visit.
  Iron is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Magnesium | 0, 3, 5 and 10 years since the selection visit.
  Magnesium is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Zinc | 0, 3, 5 and 10 years since the selection visit.
  Zinc is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Insulin | 0, 3, 5 and 10 years since the selection visit.
  Insulin is measured both in micro international units per liter and in picograms per milliliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Insulin resistance | 0, 3, 5 and 10 years since the selection visit.
  The Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) index is used to estimate insulin resistance.
Biochemical analysis: C-reactive protein | 0, 3, 5 and 10 years since the selection visit.
  C-reactive protein is measured in milligrams per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Tumor necrosis factor alpha | 0, 3, 5 and 10 years since the selection visit.
  Tumor necrosis factor alpha is measured in picograms per deciliter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Adiponectin | 0, 3, 5 and 10 years since the selection visit.
  Adiponectin is measured in milligrams per liter on an individual basis. Analysis performed in plasma.
Biochemical analysis: Energy | 0, 3, 5 and 10 years since the selection visit.
  Energy is determined in kilocalories on an individual basis. Analysis performed in plasma.
Biochemical analysis: Carbohydrates | 0, 3, 5 and 10 years since the selection visit.
  Carbohydrates are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Sugars | 0, 3, 5 and 10 years since the selection visit.
  Sugars are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Fiber | 0, 3, 5 and 10 years since the selection visit.
  Fibers are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Polysaccharides | 0, 3, 5 and 10 years since the selection visit.
  Polysaccharides are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Total fat | 0, 3, 5 and 10 years since the selection visit.
  Total fat is measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Saturated fatty acids | 0, 3, 5 and 10 years since the selection visit.
  Saturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Monounsaturated fatty acids | 0, 3, 5 and 10 years since the selection visit.
  Monounsaturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Polyunsaturated fatty acids | 0, 3, 5 and 10 years since the selection visit.
  Polyunsaturated fatty acids are measured in grams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B1 | 0, 3, 5 and 10 years since the selection visit.
  Vitamin B1 is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B2 | 0, 3, 5 and 10 years since the selection visit.
  Vitamin B2 is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B3 | 0, 3, 5 and 10 years since the selection visit.
  Vitamin B3 is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B6 | 0, 3, 5 and 10 years since the selection visit.
  Vitamin B6 is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B9 | 0, 3, 5 and 10 years since the selection visit.
  Vitamin B9 is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin B12 | 0, 3, 5 and 10 years since the selection visit.
  Vitamin B12 is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin C | 0, 3, 5 and 10 years since the selection visit.
  Vitamin C is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin A | 0, 3, 5 and 10 years since the selection visit.
  Vitamin A is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin D | 0, 3, 5 and 10 years since the selection visit.
  Vitamin D is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Vitamin E | 0, 3, 5 and 10 years since the selection visit.
  Vitamin E is measured in milligrams on an individual basis. Analysis performed in plasma.
Biochemical analysis: Carotenes | 0, 3, 5 and 10 years since the selection visit.
  Carotenes are measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Retinol | 0, 3, 5 and 10 years since the selection visit.
  Retinol is measured in micrograms on an individual basis. Analysis performed in plasma.
Biochemical analysis: Water | 0, 3, 5 and 10 years since the selection visit.
  Water is measured in grams on an individual basis. Analysis performed in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Gil, Principal Investigator — Universidad de Córdoba; Nancy E Babio, Principal Investigator — University Rovira i Virgili
Locations (8):
- Spain (8):
  - University of Santiago de Compostela, Santiago de Compostela, La Coruña
  - University of Navarra, Pamplona, Navarre
  - Institut Hospital del Mar d'Investigacions Mèdiques, Barcelona
  - University of Cordoba, Córdoba
  - University of Granada, Granada
  - Rovira i Virgili University, Tarragona
  - University of Valencia, Valencia
  - University of Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analysed during the current study are not publicly available due to data regulations and for ethical reasons, considering that this information might compromise research participants' consent because our participants only gave their consent for the use of their data by the original team of investigators. Collaboration for data analyses can be requested to estudiocoral@corals.es

REFERENCES:
- [Derived] Vazquez-Bolea N, Mora-Martinez C, Cuervo M, Martinez JA, Gil-Campos M, Leis R, Babio N, Moreno LA, Corella D, Moreira Echeverria A, Aguilera CM, Castro-Collado C, Picans-Leis R, Hernandez-Cacho A, Miguel-Berges ML, Martin-Climent P, Jurado-Castro JM, Vazquez-Cobela R, Plaza-Diaz J, Rueda-De Torre I, Pastor-Villaescusa B, de la Torre-Aguilar MJ, Salas-Salvado J, Sanz Y, Navas-Carretero S. Gut microbiota composition and derived enterotypes are associated with ponderal status in preschool children. Childhood obesity risk assessment longitudinal study (CORALS) cohort. Clin Nutr. 2026 Feb;57:106558. doi: 10.1016/j.clnu.2025.106558. Epub 2025 Dec 29. PMID 41499920
- [Derived] Jurado-Castro JM, Pastor-Villaescusa B, Castro-Collado C, Gil-Campos M, Leis R, Babio N, Moreno LA, Navas-Carretero S, Portoles O, Echeverria AM, De La Torre-Aguilar MJ, Picans-Leis R, Salas-Salvado J, de Miguel-Etayo P, Flores-Rojas K, Vazquez-Cobela R, Sales JV, Miguel-Berges ML, Izquierdo-Lopez I, Gomez-Martinez C, Cordoba-Rodriguez DP, Mimbrero G, Llorente-Cantarero FJ; CORAL Study investigators. Evaluation of Physical Activity, Sedentary Patterns, and Lifestyle Behavior in Spanish Preschool Children from the CORALS Cohort. Sports Med Open. 2025 Jun 9;11(1):71. doi: 10.1186/s40798-025-00865-2. PMID 40490568
- See also: Official website of the study. On this page you will find general information about the study, the participating teams and their contacts, as well as the latest news about the study. — https://corals.es/